CLINICAL TRIAL: NCT03734614
Title: Preventive Effects of Low-dose Aspirin as Adjuvant Therapy After Radical Nephrectomy on Disease Recurrence/Metastasis and Survival in Patients With Locally Advanced Renal Cell Carcinoma: an Observational Prospective Cohort Study
Brief Title: Preventive Effects of Aspirin as Adjuvant Therapy in Patients With Locally Advanced Renal Cell Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Yiran Huang, Professor of Urology, RenJi Hospital
Other Study IDs: RCC ASA PREVENT1
Record Dates: First submitted 2018-10-28; First posted 2018-11-08 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2018-11

CONDITIONS: Aspirin as Adjuvant Therapy in Patients With Surgically Treated High Risk Renal Cell Carcinoma
Keywords: asprin; locally advanced; renal cell carcinoma; adjuvant therapy
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Aspirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with adjuvant aspirin: After surgery, patients would use low-dose aspirin (100mg) longer than 1 year
  Interventions: Drug: Low dose of aspirin
- Patients without adjuvant aspirin: After surgery, patients would not use low-dose aspirin or use asprin shorter than 1 year

INTERVENTIONS:
Drug: Low dose of aspirin — Low dose of aspirin, 100 mg daily for longer than one year
  Groups: Patients with adjuvant aspirin

SUMMARY:
The study evaluates the protective effect of low-dose aspirin use as adjuvant therapy on locally advanced renal cell carcinoma in users and non-users of aspirin in Renji Hospital, Shanghai, China.

DETAILED DESCRIPTION:
Renal cell carcinoma (RCC) accounts for 2%~3% of all malignant tumors worldwide. In China, the incidence of renal cancer is increasing year by year. It is reported about one-third of patients were at late stage when diagnosed while about one-third of patients who received surgical treatment would eventually lead to recurrence or metastasis. The 5-years survival is only about 50% in patients with locally advanced RCC, which lacks of effective adjuvant treatments, although the S-TRAC study showed improved Disease-free Survival (DFS) in high-risk renal cell carcinoma after nephrectomy.

Aspirin, also called acetylsalicylic acid, belongs to non-steroidal anti-inflammatory drugs (NSAIDs). Its inhibitory effect on platelet aggregation makes it widely used in cardiovascular and cerebrovascular diseases. In addition, a number of epidemiology, basic and clinical researches confirmed that aspirin may be the most promising chemopreventive agent to date, especially against CRC. Prospective studies have also shown that aspirin can improve survival of patients with breast cancer,colorectal cancer, gastro-esophageal cancer and prostate cancer.

In the investigator's clinical practice, we'd like to investigate the preventive effects of low-dose aspirin use as an adjuvant therapy after radical nephrectomy on disease recurrence/metastasis and survival in patients with locally advanced renal cell carcinoma in Renji Hospital affiliated to Shanghai Jiao Tong University school of medicine. The study is observational and prospective, patients with locally advanced RCC will decide whether or not to take low-dose Aspirin(100mg/d) after radical nephrectomy as adjuvant therapy for 1 year. The primary end point was the duration of disease-free survival, and the secondary end points included overall survival and safety.

ELIGIBILITY:
Inclusion Criteria:

* Patients must complete radical surgery more than 4 weeks and less than 12 weeks prior to study entry
* Patients must have histologically or cytologically confirmed renal cell carcinoma. Using 2017 (American Joint Committee on Cancer [AJCC] 8th edition) TNM Staging, patients must be one of the following:
* pT2aG3 or G4N0M0
* pT2bG(any)N0M0
* pT3G(any)N0M0
* pT4G(any)N0M0
* pT(any)G(any)N1M0
* Patients must have no clinical or imaging evidence of visible residual lesions or distant metastases (M0) after nephrectomy
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Patients must be able to swallow pills

Exclusion Criteria:

* Patients with haemorrhagic diathesis (i.e. haemophilia).
* Patients with prior malignant tumors except for kidney cancers in the past 5 years.
* Patients with documented or suspected metastases.
* Patients with serious, nonhealing wound, ulcer, or bone fracture.
* Patients with a history of stroke, coronary arterial disease, angina, or vascular disease.
* Patients who are pregnant, lactating, or not using adequate contraception.
* Patients who have known allergy to NSAID or Aspirin.
* Patients receiving other antiplatelet agents (i.e. clopidogrel, ticlopidine) or anticoagulants (i.e. warfarin, low molecular weight heparins).
* Patients receiving current long term treatment (≥1 month) with Aspirin or other NSAIDs.
* Subject unwilling or unable to comply with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with locally advanced renal cell carcinoma undergoing radical nephrectomy
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2018-10-08 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Disease-free Survival | 36 mouths
  Disease-free Survival

SECONDARY OUTCOMES:
Overall survival | 36 months
  Overall survival
Cancer specific survival | 36 months
  Cancer specific survival
adverse event rate | 12 months
  Rate of patients with each of the adverse event per grade

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No